CLINICAL TRIAL: NCT01938950
Title: Resistance and Cardiorespiratory Time-matched Exercise in Youth: A Randomized Clinical Trial (RCT:RCT)
Acronym: RCT:RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the institution
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, SoJung Lee, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO12080401; 1R01HL114857-01A1 (NIH)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Aerobic Exercise (Active Comparator): Participants will perform aerobic exercise using treadmills and/or ellipticals at 40-65% of VO2peak, three times per week, for 60 minutes/session.
  Interventions: Other: Aerobic Exercise
- Resistance Exercise (Active Comparator): Participants will perform 2 sets (8-12 repetitions per set) of 8 exercises to the point of failure using weight stack equipment, three times per week, for 60 minutes/session. 2 sets of push-ups and sit-ups will also be performed.
  Interventions: Other: Resistance Exercise
- Aerobic and Resistance Exercise (Active Comparator): Participants will perform aerobic exercise using treadmills and/or ellipticals for 30 min at 40-65% of VO2peak and thereafter, perform 1 set of each of the above 10 resistance exercise for 30 min.
  Interventions: Other: Aerobic and Resistance Exercise

INTERVENTIONS:
Other: Aerobic Exercise
  Arms: Aerobic Exercise
Other: Resistance Exercise
  Arms: Resistance Exercise
Other: Aerobic and Resistance Exercise
  Arms: Aerobic and Resistance Exercise

SUMMARY:
The current epidemic rate of childhood obesity is a leading health concern as overweight/obese youth may suffer from comorbid conditions, once considered exclusive to adults. It has been suggested that physical inactivity is a major determinant of obesity and obesity-related health risk in children and adolescents. Recent studies in adults report that the combination of aerobic and resistance exercise is a better strategy than aerobic or resistance exercise alone for reducing risk factors for type 2 diabetes. Currently, the most effective exercise modality for concurrent reductions of adiposity, in particular abdominal fat, and risk factors for type 2 diabetes and cardiovascular disease (CVD) is unknown in adolescents. Therefore, we will employ a randomized trial to examine the effects of a long-term aerobic exercise, resistance exercise, and a combination of both exercise regimens on: 1) in vivo insulin sensitivity, glucose tolerance and risk for type 2 diabetes, 2) total adiposity, skeletal muscle mass, visceral adiposity and ectopic fat in the liver and skeletal muscle, and 3) traditional and non-traditional risk factors/markers for CVD in overweight boys and girls. We will recruit 168 sedentary overweight (BMI >85th percentile) adolescent boys and girls aged 12-17 years old and randomly assign them to one of three 6-month intervention groups (n = 56 each group): 1) aerobic exercise (180 min/week), 2) resistance exercise (180 min/week), or 3) aerobic and resistance exercise (180 min/week) group. A weight maintenance diet (55-60% carbohydrate, 15-20% protein, and 25-30% fat) will be prescribed and monitored for all groups, so that any changes in energy balance will be induced by exercise intervention alone (e.g., no calorie restriction). We believe that this proposed application will have a significant implication that is directly relevant for one in three American adolescents who are at increased risk of developing obesity-related co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

Age 12-17 years

* BMI percentile for age and sex >-85% percentile and BMI <40 kg/m2
* No structured physical activity in the past 3 months prior to the study (not including school physical education classes)
* No significant weight changes (>2-3 kg/m2) in the past 3 months prior to the study

Exclusion Criteria:

* Endocrine disorders (e.g., polycystic ovary syndrome, diabetes)
* Syndromic obesity
* Positive pregnancy test
* Use of chronic medications which influence glucose metabolism and body composition
* Chronic medical/psychiatric conditions preventing the ability to participate in the study.
* Anemia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 6 months

SECONDARY OUTCOMES:
Total and regional body composition | 6 months
  Total fat, visceral fat, intrahepatic lipid, skeletal muscle lipid, skeletal muscle mass
Cardiovascular disease risk factors | 6 months
  Carotid intima-media thickness, arterial stiffness, endothelial dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: SoJung Lee, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Yu WW, Lee S, Arslanian S, Tamim H, Kuk JL. Effects of Exercise on Resting Metabolic Rate in Adolescents with Overweight and Obesity. Child Obes. 2021 Jun;17(4):249-256. doi: 10.1089/chi.2020.0280. Epub 2021 Mar 18. PMID 33739874
- [Derived] Kuk JL, Lee S. Assessing the utility of cardiorespiratory fitness, visceral fat, and liver fat in predicting changes in insulin sensitivity beyond simple changes in body weight after exercise training in adolescents. Appl Physiol Nutr Metab. 2021 Jan;46(1):55-62. doi: 10.1139/apnm-2020-0284. Epub 2020 Jul 16. PMID 32674604
- [Derived] Lee S, Libman I, Hughan KS, Kuk JL, Barinas-Mitchell E, Chung H, Arslanian S. Effects of exercise modality on body composition and cardiovascular disease risk factors in adolescents with obesity: a randomized clinical trial. Appl Physiol Nutr Metab. 2020 Dec;45(12):1377-1386. doi: 10.1139/apnm-2019-0993. PMID 32674587
- [Derived] Kuk JL, Lee S. Sex and Ethnic Differences in the Relationship between Changes in Anthropometric Measurements and Visceral Fat in Adolescents with Obesity. J Pediatr. 2019 Oct;213:121-127. doi: 10.1016/j.jpeds.2019.05.052. Epub 2019 Jun 22. PMID 31235380
- [Derived] Lee S, Libman I, Hughan K, Kuk JL, Jeong JH, Zhang D, Arslanian S. Effects of Exercise Modality on Insulin Resistance and Ectopic Fat in Adolescents with Overweight and Obesity: A Randomized Clinical Trial. J Pediatr. 2019 Mar;206:91-98.e1. doi: 10.1016/j.jpeds.2018.10.059. Epub 2018 Dec 13. PMID 30554789